CLINICAL TRIAL: NCT05061160
Title: Acute Effects of Continuous Verses Interval Aerobic Training on Autonomic Dysreflexia in Spinal Cord Injury Patient
Brief Title: Acute Effects of Continuous Verses Interval Aerobic Training in Spinal Cord Injury Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01080 Maryam Tahir
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
Keywords: Continuous Aerobic Exercise; Interval Aerobic Exercise
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval Aerobic Exercise training Group (Experimental): Interval Aerobic Exercise for 4 weeks
  Interventions: Other: Interval Aerobic Exercise training Group
- Continuous Aerobic Exercise training Group (Active Comparator): Continuous aerobic exercise for 4 weeks
  Interventions: Other: Continuous Aerobic Exercise training Group

INTERVENTIONS:
Other: Interval Aerobic Exercise training Group — Interval Aerobic exercise will be on upper limb Bicycle with a pause of 3 mins interval Interval Aerobic Exercises: Frequency= 3 times per week Intensity= 50% of heart rate reserve for 2 mins 80% of heart rate reserve for 1 min Type= interval aerobic exercise Time= 40 minutes
  There will be 5 minutes for warm up and 5 minutes for cool down.
  Arms: Interval Aerobic Exercise training Group
Other: Continuous Aerobic Exercise training Group — Continuous Aerobic exercise will be on upper limb Bicycle Continuous Aerobic Exercise: Frequency= 3 times per week Intensity= 50% of heart rate reserve Type= continuous aerobic exercise Time= 40 minutes
  There will be 5 minutes for warm up and 5 minutes for cool down.
  Arms: Continuous Aerobic Exercise training Group

SUMMARY:
To determine the Acute effects of continuous verses interval aerobic training on autonomic dysreflexia in Spinal Cord injury Patient. To Determine the Acute effects of these training on, Exercise Self efficacy and pain.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury Patients with level of injury below T 10
* Acute Spinal Cord Injury (Usually Acute phase lasts 8-12 weeks)
* Patients Had experience of Syncope or Postural Hypotension

Exclusion Criteria:

* Neurological disease,
* Cognitive impairment (Mini-Mental State Examination < 22) ,
* Acute and chronic infections

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Baroreflex sensitivity (BRS) | 4th Week
  BRS is the index which is used to quantify the control of baroreflex on the heart rate. Patient's beat to beat arterial pressure and heart rate are measured simultaneously with the Maximal expiratory pressure (MEP) manoeuvre or valsalva manoeuvre. Changes from the baseline to 4 week will be analyzed
Heart rate reserve (HRR) | 4th Week
  It is the difference between resting heart rate and maximum heart rate. HRR is primarily use to determine heart rate zone for exercise. HRR can be calculated by subtracting resting heart rate from maximum heart rate. Changes from the baseline to 4 week will be analyzed
Systolic and diastolic blood pressure | 4th week
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer

SECONDARY OUTCOMES:
Oxygen saturation | 4th Week
  Amount of oxygen in the blood is known as oxygen saturation. normal range is 94-99 percent. Pulse oximeter is used to measure oxygen saturation. Changes from the baseline to 4 weeks
Pain perception | 4th week
  Pain is defined as unpleasant sensation which is generated by body as a protective response to prevent further tissue damage. It will be measured with the help of Numeric pain rating scale ranging 0 to 10. where 0 is no pain and 10 is the worst pain imaginable. Changes from the baseline to 4 week will be analyzed
Exercise self-efficacy | 4th week
  It is defined as how much an individual consider he eligible to perform the given exercise. Spinal Cord Injury (SCI) Exercise Self Efficacy scale will be provided to the individuals at the baseline and then after 72 hours i.e 3 days of training/week. It has total of 10 questions which allow the participants to indicate on four point scale how much confident they are about the exercise.
QOL Index-Spinal cord injury version questionnaire | 4th Week
  QOL index spinal cord injury version is used to assess the quality of life of spinal cord injury patients. It has 32 to 37 items. Each item is rated on scale of 1 to 6.5 scores of 0-30 are calculated.1) quality of life, 2) health and functioning, 3) social and economic life, 4) physiological life, and 5) family life. Changes from the baseline to 4th week will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Armed Forces Institute of Rehabilitation Sciences, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No